CLINICAL TRIAL: NCT05112432
Title: EPI-MINN: Targeting Cognition and Motivation in Coordinated Specialty Care for Early Psychosis
Brief Title: EPI-MINN: Targeting Cognition and Motivation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSYCH-2021-30030; Pro00049491 (Other: Advarra IRB); 1R01MH120589 (NIH)
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Psychosis
Keywords: Cognitive Training; Motivation Enhancement; First Episode Psychosis; Schizophrenia Spectrum Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — PRIME protocol; Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment as Usual (Active Comparator): Participants will be treated as usual and will not complete cognitive training or use the Personalized Real-Time Motivational Enhancement App. Participants may choose to complete study activities in person at their coordinated specialty care program or may choose to complete study activities remotely.
  Interventions: Other: Early Psychosis Coordinated Specialty Care
- Cognitive Training plus Personalized Real-Time Intervention for Motivational Enhancement App (PRIME) (Experimental): The Mobile Intervention. 20 hours of training consisting of 10 hours of cognitive training exercises plus 10 hours of social cognitive training exercises will be delivered over the course of 12 weeks in addition to PRIME. Participants may choose to complete study activities in person at their coordinated specialty care program or may choose to complete study activities remotely.
  Interventions: Device: Cognitive and Social Cognitive Training; Behavioral: Personalized Real-Time Intervention for Motivational Enhancement (PRIME) App; Other: Early Psychosis Coordinated Specialty Care

INTERVENTIONS:
Device: Cognitive and Social Cognitive Training — The Cognitive Training Module is designed to improve the speed and accuracy of auditory information processing while engaging working memory and cognitive control under conditions of close attention and reward. Exercises continuously adjust difficulty level to user performance to maintain an approximately 80% current performance rate. The goal is to increase the effectiveness by which salient stimuli engage and drive plastic changes in brain systems that in individuals with psychosis exhibit relatively poor temporal response.
  The Social Cognition Training Module consists of exercises designed to ameliorate core deficits in social cognition expressed in schizophrenia and Autism Spectrum Disorders. The exercises apply principles of implicit learning to restore the brain's capacity to process and utilize socially-relevant information, and include training to improve affect perception, social cue perception, theory of mind, self-referential style, and emotion labeling and working memory.
  Arms: Cognitive Training plus Personalized Real-Time Intervention for Motivational Enhancement App (PRIME)
Behavioral: Personalized Real-Time Intervention for Motivational Enhancement (PRIME) App — The PRIME smartphone-based app is designed to be used for 12 weeks to enhance motivation in people with early psychosis. Participants work towards self-identified goals with the support of the virtual community of age-matched peers, as well as with motivation coaches. Participants discuss their interests and aspirations with each other and with their coach, and the coach sends daily individualized motivational messages. Coaches also provide tailored interventions to enhance motivation, and post daily discussion topics to the PRIME community to encourage interaction between members. Coaches will maintain close communication and feedback on progress with each individual's clinical team.
  Arms: Cognitive Training plus Personalized Real-Time Intervention for Motivational Enhancement App (PRIME)
Other: Early Psychosis Coordinated Specialty Care — Participants will continue to receive treatment as usual at their early psychosis coordinated specialty care clinics. These clinics may follow the NAVIGATE model, as an example.

SUMMARY:
The purpose of this study is to perform a practice-based research project designed to assess whether cognition and motivated behavior in early psychosis can be addressed as key treatment goals within real-world settings by using a 12-week mobile intervention program. Participants who are enrolled in a chart review study of measurement-based care will be recruited to participate in this study. In the measurement-based care study, participants are enrolled in coordinated specialty care programs for early psychosis that provide comprehensive clinical services such as psychotherapy, medication management, psychoeducation, work or education support, and measurement-based care. Participants will complete a set of well-defined measures every 6 months that assess symptoms, functioning, cognition and motivation as standard of care. The current study will utilize the data acquired in the measurement-based care study.

The aim of this study is to investigate a well-defined 12-week mobile intervention program specifically designed to target cognitive functioning and motivated behavior for individuals with early psychosis. The investigators will test for differences in the clinical trajectories over 18 months in those who receive the intervention vs. those who do not.

This study will be conducted jointly with a sister protocol under a separate NCT listing. This iteration will be conducted locally within the EPI-MINN Network, while the other project will be conducted on a national scale.

DETAILED DESCRIPTION:
Cognitive dysfunction is a core pathophysiological feature of psychosis and one of the strongest predictors of functional outcomes. Several studies indicate that current early intervention programs may not significantly alter long-term clinical outcome, suggesting that critical treatment target(s), beyond symptoms and functional status, are not being addressed. Evidence strongly indicates that, along with cognitive dysfunction, impaired motivation is also a critical target and unmet therapeutic need.

The application of effective treatment to improve cognition in early phases of psychosis has a very high likelihood of significantly improving long-term community functioning. The investigators have demonstrated both behavioral gains and improved neural system functioning after neuroscience-informed cognitive training in schizophrenia, in both chronic and early phases of the illness. In young recent-onset individuals (average age of 21 years), the investigators' multi-site double-blind randomized controlled trial showed that 40 hours/ 10 weeks of cognitive training delivered at home over a laptop resulted in significant gains in global cognition, verbal memory, and problem solving compared to a computer games control condition. Cognitive gains were significantly correlated with enhanced thalamic volume and thalamo-cortical connectivity, as well as increased white matter integrity. A meta-analysis of 11 RCTs in early schizophrenia has also indicated the benefit of cognitive remediation approaches.

Impaired motivation is also a core feature and very strong predictor of functional outcome in early stages of psychosis. Some studies have shown positive effects in improving motivation immediately after the intervention, but treatments that induce enduring improvements in motivated behavior are scarce. Disturbances in motivated behavior reflect a range of factors, including diminished anticipatory pleasure, difficulty learning from rewarding outcomes, reduction in effort expended to obtain rewarding outcomes, and impairment and disconnection between components of social motivation. This makes it difficult to determine optimal therapeutic approaches. However, some headway is starting to appear in the literature. For instance, social cognition impairments appear to play a specific contributing role to dysfunctions in motivated behavior, and are amenable to intervention. We have found that ratings of motivated behavior improve after social cognition training, and are significantly greater in subjects who performed cognitive training combined with social cognition training, than in those who completed only cognitive training. The investigators have also demonstrated a significant relationship between 6-month social functioning and training-induced improvements in the neural correlates of a self-other reality monitoring task. These data, along with the literature on reward anticipation and on social engagement in psychosis, led this group to work with young clients in a user-centered design process, to develop a mobile app called Personalized Real-time Intervention for Motivational Enhancement (PRIME). The app has been extremely well received by users and published behavioral findings are highly promising. Thus, the investigators will combine a focused course of cognitive plus social cognitive training (delivered remotely) with PRIME, to address the cognitive dysfunction and impaired motivation.

Functional recovery lags behind symptom recovery in early intervention programs, is sometimes difficult for individuals to attain, and is closely aligned with cognitive and motivational deficits. How could outcomes for individuals with early psychosis to improved? The results from the EPI-MINN: Measurement-Based Care study will provide data-driven knowledge on factors that contribute to 2-year treatment response trajectories in early psychosis. This knowledge will be combined with insights from the investigators' current study to deepen understanding of methods to optimize coordinated specialty care to improve clinical trajectories, using a well-defined scalable mobile program that addresses as-of-yet unmet therapeutic needs.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in EPI-MINN: Measurement Based Care protocol, STUDY00009334
* Good general health (i.e. not acutely ill or experiencing a severe/chronic illness that would impede their ability to complete study activities. This determination shall be, if necessary, made at the discretion of the PIs)
* Estimated IQ at or above 70, as estimated by the Penn CNP Matrix Reasoning Test
* Achieved clinical stability, defined as outpatient status for at least one month prior to study participation and clinically stable doses of psychiatric medication (by PI discretion) for at least one month prior to study participation (including no medication)
* Has access to a smartphone or other mobile device to use the PRIME app

Exclusion Criteria:

* Under legal commitment to treatment or is under medical guardianship, and there is no provision in the guardianship order or a court order to allow the guardian to consent to participation in research
* Participated in significant cognitive training programs within the last three years
* Diagnosed with a neurological disorder (Autism Spectrum Disorder is allowed)
* Clinically significant substance abuse that is impeding the participant's abulity to participate fully during recruitment, enrollment, assessment, or training, (is unable to remain sober for assessments and training)
* Risk of suicidal behavior, as indicated by the clinicall obtained C-SSRS or clinician judgement. Risk of suicidal behavior is defined as:

  * Active suicidal ideation at screening or baseline, or
  * Previous intent to act on suicidal ideation with a specific plan, preparatory acts, or an actual suicide attempt within the last 3 months

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change Penn Computerized Neuropsychological Testing System (Penn CNP) Scores | 18 months
  Penn CNP is reported as the total score on 4 cognitive domains. The DSST ranges from 0-300+, the PWMT ranges from 0-40, the PMAT ranges from 0-24, and the ER-40 ranges from 0-40. Penn CNP will be assessed at baseline, during pre-training, at 6 months, 12 months, and 18 months. Higher accuracy scores indicate higher cognitive function and lower reaction time scores indicate faster reaction time. Reaction time is reported in milliseconds. Performance score is calculated based on accuracy and reaction speed.
Change in Test My Brain Scores | 18 months
  Test My Brain is reported as the total score on 4 cognitive domains. The Digit Symbol Matching ranges from 0 -300+, the Verbal Paired Associated ranges from 0 - 25, the Matrix Reasoning ranges from 0 - 35, and the Multiracial Face Emotion Identification Test ranges from 0 - 48. Test My Brain will be assessed at baseline, during pre-training, at 6 months, 12 months, and 18 months. Higher scores indicate higher cognitive function. Performance score is calculated based on accuracy and reaction speed.
Change in Dysfunctional Attitudes Scale - Defeatist Beliefs Subscale (DAS-DB) Score | 18 months
  DAS-DB is measured over 14 items with total scores ranging from 14-98, where higher scores indicate greater defeatist beliefs. DAS-DB will be assessed at baseline, 6 months, 12 months, and 18 months.
Quality of Life Scale - Abbreviated | 18 months
  The quality of life scale contains 9 items rated from 0 to 6, with higher scores indicating increased functioning/decreased symptom severity. Outcome is reported as 9 separate domain scores.
Change in Behavioral Inhibition and Activation Scale (BIS/BAS) - BIS Score | 18 months
  BIS/BAS BIS questionnaire consists of 24 items with total scores ranging from 7-28, where higher scores indicate greater sensitivity to negative aspects of goals. BIS/BAS BIS will be assessed at baseline, 6 months, 12 months, and 18 months.
Change in Behavioral Inhibition and Activation Scale (BIS/BAS) - BAS Reward Responsiveness Score | 18 months
  BIS/BAS BAS reward responsiveness questionnaire consists of 24 items with total scores ranging from 5-20, where higher scores indicate greater tendency to be influenced by the possibility of reward when pursuing a goal. BIS/BAS BAS reward responsiveness will be assessed at baseline, 6 months, 12 months, and 18 months.
Change in Behavioral Inhibition and Activation Scale (BIS/BAS) - BAS Drive Score | 18 months
  BIS/BAS BAS drive questionnaire consists of 24 items with total scores ranging from 4-16, where higher scores indicate greater persistence in efforts towards obtaining a goal. BIS/BAS BAS drive will be assessed at baseline, 6 months, 12 months, and 18 months.
Change in Behavioral Inhibition and Activation Scale (BIS/BAS) - BAS Fun Seeking Score | 18 months
  BIS/BAS BAS fun seeking questionnaire consists of 24 items with total scores ranging from 4-16, where higher scores indicate greater tendency to be influenced by novelty and seeking out new experiences. BIS/BAS BAS fun seeking will be assessed at baseline, 6 months, 12 months, and 18 months.
Change in Motivation and Pleasure Scale - Self Report (MAPS-SR) - Social Pleasure Score | 18 months
  MAPS-SR social pleasure questionnaire consists of 15 items with total scores ranging from 0-12, where higher scores indicate increased pathology in this domain. MAPS-SR social pleasure will be assessed at baseline, 6 months, 12 months, and 18 months.
Change in Motivation and Pleasure Scale - Self Report (MAPS-SR) - Recreational or Work Pleasure Score | 18 months
  MAPS-SR recreational or work pleasure questionnaire consists of 15 items with total scores ranging from 0-12, where higher scores indicate increased pathology in this domain. MAPS-SR recreational or work pleasure will be assessed at baseline, 6 months, 12 months, and 18 months.
Change in Motivation and Pleasure Scale - Self Report (MAPS-SR) - Feelings and Motivations About Close, Caring Relationships Score | 18 months
  MAPS-SR feelings and motivations about close, caring relationships questionnaire consists of 15 items with total scores ranging from 0-24, where higher scores indicate increased pathology in this domain. MAPS-SR feelings and motivations about close, caring relationships will be assessed at baseline, 6 months, 12 months, and 18 months.
Change in Motivation and Pleasure Scale - Self Report (MAPS-SR) - Motivation and Effort to Engage in Activities Score | 18 months
  MAPS-SR motivation and effort to engage in activities questionnaire consists of 15 items with total scores ranging from 0-24, where higher scores indicate increased pathology in this domain. MAPS-SR motivation and effort to engage in activities will be assessed at baseline, 6 months, 12 months, and 18 months.

SECONDARY OUTCOMES:
COMPASS-10 | 18 months
  The Compass-10 scale consists of 10 items rated on a scale from 0 to 6, with higher scores indicating more severe symptoms of depression and anxiety. Outcome will be reported as 10 separate domain scores.

OTHER OUTCOMES:
BrainHQ Cognitive Training Performance Data | 12 weeks
  The number of hours of training completed will be reported ranging from 0-20.
Tolerability of BrainHQ Cognitive Training & PRIME | 12 weeks
  This measure contains both qualitative and quantitative information. Participants will compete questionnaires regarding the tolerability for PRIME and the tolerability of BrainHQ cognitive training. A global score will be calculated and participants are categorized as low tolerability, medium tolerability, or high tolerability. Outcome will be reported as the number of participants in each tolerability category - low, medium, and high.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota Department of Psychiatry and Behavioral Sciences
Locations (3):
- United States (3):
  - Human Development Center, Duluth, Minnesota
  - Hennepin Healthcare, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota